CLINICAL TRIAL: NCT06658210
Title: Combined Effects of Soft Tissue Mobilization and Pelvic Floor Muscle Exercises on Pain, Sexual Life Quality and Functional Mobility in Women With Post-operative Adhesions After Hysterectomy
Brief Title: Effects of Soft Tissue Mobilization and Pelvic Floor Muscle Exercises on Pelvic Adhesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hunaida Iftikhar
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Pelvic Adhesions; Post Hysterectomy Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- soft tissue mobilization with pelvic floor muscle exercises (Experimental): soft tissue mobilization with pelvic floor muscle exercises
  Interventions: Other: soft tissue mobilization with pelvic floor muscle exercises
- soft tissue mobilization without pelvic floor muscle exercises (Experimental): soft tissue mobilization without pelvic floor muscle exercises
  Interventions: Other: soft tissue mobilization without pelvic floor muscle exercises

INTERVENTIONS:
Other: soft tissue mobilization with pelvic floor muscle exercises — Group A will receive soft tissue mobilization and pelvic floor muscle exercises. Soft tissue mobilization technique will include abdominal myofascial release/trigger point release and deep scar mobilization to decrease pain and improve scar mobility
  Arms: soft tissue mobilization with pelvic floor muscle exercises
Other: soft tissue mobilization without pelvic floor muscle exercises — Group B will receive soft tissue mobilization technique without pelvic floor exercises.
  Arms: soft tissue mobilization without pelvic floor muscle exercises

SUMMARY:
Adhesions are permanent tissue connections that are created by fibrin deposition between different tissue planes or organs. They are a part of the internal healing process and inflammatory reactions that go through several overlapping phases, including the proliferative phase, remodeling phase, and hemostasis/inflammatory phase. Adhesions are typically the body's defense mechanisms against various triggers of inflammation, including physical, chemical, and infections. These triggers can have unfavorable consequences, including chronic pain, obstruction (particularly bowel), functional impairment, and infertility. This may cause adjacent structures to lose their flexibility and mobility. The nonsurgical treatment of symptoms thought to be associated with adhesions has centered on several methods of soft tissue scar removal.

DETAILED DESCRIPTION:
This study will be randomized controlled trial and will be conducted in Hanif medical center and poly clinic and Lady willingdon hospital. The total duration of treatment will be 10 week.

Non-probability convenience sampling technique will be used and 56 participants will be recruited in study after randomization. The subjects will be divided into two groups. Group A will receive soft tissue mobilization of pelvic area with pelvic floor muscle exercises and Group B will receive soft tissue mobilization of pelvic area without pelvic floor muscle exercises after heating for 10 minutes as baseline treatment. The tools that will be used are Numeric Pain Rating Scale (NPRS), Female Sexual Function Index (FSFI) and Functional status questionnaire (FSQ). After data collection data will be analyzed by using SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Married women
* Age 40-60 years
* BMI below 30 (13)
* Women with post-operative pelvic adhesions (14)
* Women after hysterectomy (3 months after surgery)

Exclusion Criteria:

* Women with any other surgery
* Women with failed pelvic surgery (14)
* Post-operative women with open wound (unhealed suture site) (14)
* Women with uncontrolled hypertension, thrombophlebitis, hematoma, osteomyelitis, myositis ossificans and malignancy

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 56 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | 6 weeks
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.
Female sexual function index | 6 weeks
  The FSFI questionnaire consists of 19 close-ended questions related to sexual activity and includes six domains:
  * Sexual desire (question number 1-2)
  * Sexual arousal (question number 3-6)
  * Lubrication (question number 7-10)
  * Orgasm (question number 11-13)
  * Sexual satisfaction (question number 14-19)
Functional status questionnaire | 6 weeks
  The Functional Status Questionnaire (FSQ) is a brief, self-administered questionnaire developed by researchers from Boston's Beth Israel Hospital and the University of California at Los Angeles. The FSQ was designed to screen for disability and to monitor clinically meaningful change in function.

CONTACTS AND LOCATIONS:
Overall Officials: Hunaida Iftikhar Hunaida Iftikhar, MSPT*, Principal Investigator — Riphah International University
Locations (1):
- Hanif Medical centre and Polyclinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lang J, Ma D, Xiang Y, Hua K, Liu K, Pan L, Wang P, Yao S, Zhao F, Cheng W, Cui M, Guo H, Guo R, Hong L, Li P, Liu M, Meng Y, Wang H, Wang J, Wang W, Wu M, Yang X, Zhang J. Chinese expert consensus on the prevention of abdominal pelvic adhesions after gynecological tumor surgeries. Ann Transl Med. 2020 Feb;8(4):79. doi: 10.21037/atm.2020.02.53. PMID 32175372
- [Background] Hu Q, Xia X, Kang X, Song P, Liu Z, Wang M, Lu X, Guan W, Liu S. A review of physiological and cellular mechanisms underlying fibrotic postoperative adhesion. Int J Biol Sci. 2021 Jan 1;17(1):298-306. doi: 10.7150/ijbs.54403. eCollection 2021. PMID 33390851
- [Background] Li YT, Liu CH, Wang PH. Pelvic adhesion: A challenge of all gynecologic surgeries. J Chin Med Assoc. 2022 Aug 1;85(8):813-814. doi: 10.1097/JCMA.0000000000000756. Epub 2022 Aug 19. No abstract available. PMID 35648144